CLINICAL TRIAL: NCT02618018
Title: An Investigator-Initiated Trials on the Efficacy and Stability of AT TORBI 709M 4-haptic Toric IOL in Cataract Surgery
Brief Title: Clinical Evaluation of Efficacy and Stability of AT TORBI 709M 4-haptic Toric IOL in Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT TORBI 709M toric IOL
Record Dates: First submitted 2015-05-20; First posted 2015-12-01 (Estimated); Last update posted 2015-12-01 (Estimated); Status verified 2015-11

CONDITIONS: Iol; Astigmatism
Keywords: astigmatism; toric intraocular lens
MeSH Terms: conditions — Intraocular Lymphoma; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intraocular lens (Experimental): AT TORBI 709M toric intraocular lens
  Interventions: Procedure: AT TORBI 709M

INTERVENTIONS:
Procedure: AT TORBI 709M — Cataract surgery with AT TORBI 709M 4-haptic toric IOL

SUMMARY:
The purpose of this study is to evaluate the efficacy and stability of AT TORBI 709M 4-haptic toric IOL in cataract surgery.

DETAILED DESCRIPTION:
Inclusion criteria

1. senile cataract
2. patients' age of 21 years or older
3. preoperative regular corneal astigmatism between 1.00 D and 6.00 D

Exclusion criteria

1. pregnant, lactating women
2. presence of other ocular diseases which affect stability of lens capsule

Primary outcome : efficacy index (visual acuity, refractive results Secondary outcome : rotational stability, endothelial cell count, cornea thickness

ELIGIBILITY:
Inclusion Criteria:

* senile cataract
* patients' age of 21 years or older
* preoperative regular corneal astigmatism between 1.00 D and 6.00 D

Exclusion Criteria:

* pregnant, lactating women
* presence of other ocular diseases which affect stability of lens capsule

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Visual acuity, refractive results | 3 months
  uncorrected distance visual acuity (UCDVA) and best corrected distance visual acuity (BCDVA) measured using logarithm of the minimum angle of resolution (logMAR) refractive results measured by keratometry

SECONDARY OUTCOMES:
Rotational stability | 3 months
  Photographic evaluation of IOL rotation using slit-lamp digital photographs at each postoperative visit, and determine changes in the lens axis between visits.
Endothelial cell count | 3 months
  measured by specular microscopy
Cornea thickness | 3 months
  measured by ultrasound pachymetry

CONTACTS AND LOCATIONS:
Overall Officials: Mee Kum Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea